CLINICAL TRIAL: NCT04102215
Title: The Efficacy of a Minimally Invasive Direct Cochlear Access Via the HEARO Procedure
Acronym: ARCI25
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Vedat Topsakal (Other)
Responsible Party: Sponsor-Investigator, Prof. Vedat Topsakal, Principal Investigator, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000523
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: SIngle arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARCI25 (Experimental): Robot assited Cochlear implant surgery.
  Interventions: Device: HEARO; Device: OTOPLAN

INTERVENTIONS:
Device: HEARO — Robotic system for otological procedures
  Other Names: HEARO procedures
Device: OTOPLAN — Otological surgical planning software

SUMMARY:
To study the efficacy of a minimally invasive direct cochlear access via the HEARO procedure.

ELIGIBILITY:
Inclusion Criteria:

Adult cochlear implant candidates with suitable anatomy opting for a MED-EL cochlear implant.

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Distance of the planned trajectory to the facial nerve is < 0.4mm
* Distance of the planned trajectory to the chorda tympani is < 0.3mm
* Vulnerability
* Invalid or withdrawn informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-11-04 (Estimated)

PRIMARY OUTCOMES:
The relative ratio of the electrode array insertion into the cochlea through the drilled direct cochlea access with HEARO procedure. (Efficacy) | Image data aquired during the procedure
  The ratio of the number of the procedures in which it was possible to insert the electrode inside the cochlea through the direct cochlear access compared to the number of procedures in which the insertion through the direct cochlea access was not possible will be calculated. Aborted or converted procedures count as procedure in which insertion through the direct cochlea access was not possible. The results will be expressed in relative numbers (n of 25) and in percentage (%).

SECONDARY OUTCOMES:
Electrode array insertion depth (Efficacy) | The procedure (day 0)
  The electrode insertion depth will be measured in the post-operative image. (Degrees °)
Number of correctlly inserted electrode contact (Efficacy) | The procedure (day 0)
  The number of inserted electrode contacts into the inner ear will be counted in the post-operative image. (Number n)
  * number of contacts inserted (n)
Insertion depth prediction accuracy (Efficacy) | The procedure (day 0)
  The insertion depth prediction accuracy as the difference between the estimated insertion depth of the electrode at the planning and the actual insertion depth. (Degrees °)
Absolute angular accuracy of the drilled tunnel access | The procedure (day 0)
  The absolute in-plane and out-plane accuracy of the drilled tunnel is measured as the angular deviation between the planned and the actual angles.
Absolute lateral drilling accuracy of the drilled tunnel at the level of facial recess (Safety) | The procedure (day 0)
  The absolute lateral accuracy of the drilled tunnel to the facial nerve and chorda tympani is measured as the difference between the planned and the actual distance. (mm)
Absolute lateral drilling accuracy of the drilled tunnel at the target (Safety) | The procedure (day 0)
  The absolute lateral accuracy of the drilled tunnel is measured as the distance between the planned and actual target position. (mm)
Evaluation of the automatic landmark detection (Performance) | The procedure (day 0)
  The relative ratio of the automatically identified landmarks by OTOPLAN that were not manually adjusted by the surgeon. The intended landmarks are:
  * Middle ear cavity breakthrough
  * Bony overhang lateral wall
  * Bony overhang medial wall The absolute distance between the new position of the adjusted landmark to the position of the automatically identified landmark will be evaluated. (Number n)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Belgium

REFERENCES:
- [Derived] Heuninck E, Van de Heyning P, Van Rompaey V, Mertens G, Topsakal V. Audiological outcomes of robot-assisted cochlear implant surgery. Eur Arch Otorhinolaryngol. 2023 Oct;280(10):4433-4444. doi: 10.1007/s00405-023-07961-7. Epub 2023 Apr 12. PMID 37043021
- [Derived] Topsakal V, Heuninck E, Matulic M, Tekin AM, Mertens G, Van Rompaey V, Galeazzi P, Zoka-Assadi M, van de Heyning P. First Study in Men Evaluating a Surgical Robotic Tool Providing Autonomous Inner Ear Access for Cochlear Implantation. Front Neurol. 2022 Mar 21;13:804507. doi: 10.3389/fneur.2022.804507. eCollection 2022. PMID 35386404